CLINICAL TRIAL: NCT02279212
Title: Neuropathic Pain and Quality of Life in ICU Survivors
Acronym: NEUPAQ
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anne Kathrine Langerud, MNSc, Oslo University Hospital
Other Study IDs: S-07505b (REK)
Record Dates: First submitted 2010-12-06; First posted 2014-10-31 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Critical Illness
Keywords: Critical illness; pain; quality of life
MeSH Terms: conditions — Critical Illness; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Previous research on intensive care unit (ICU) survivors shows that rehabilitation is challenging, because of patients experiences of disease related problems both under and after treatment. Approximately 20 % of patients die within hospital, up to 80% suffer from hallucinations and nightmares, deal with paranoiac experiences, chronic pain and other symptoms and disability (Angus et al 2004; De Letter et al 2001; Ely et al 2001; Nelson et al 2006; Van den Berghe et al 2001; Van den Berghe et al 2003) . A recent study shows that 28% of intensive care survivors have chronic pain that reduce their health related quality of life (Boyle et al 2004).

The aim of this study is to perform a survey about prevalence of pain type, and which consequences this causes when it comes to function and quality of life up to 12 months after the ICU stay.

1. What type of pain has ICU survivors and how do pain change over time, related to treatment/rehabilitation and the illness' development?
2. What is the relationship between different pain characteristic, quality of life, anxiety, depression, fatigue, sleep and PTSD in these patients?
3. What is these patients largest obstacle for good QoL after discharge from hospital?

DETAILED DESCRIPTION:
A prospective and longitudinal survey 3 time points for data collection:

1. ICU - background data about the patients ICU stay (days on ventilator, medication, treatment, SAPS II, SOFA etc).
2. 3 months after ICU discharge - survey about pain, QoL, sleep, fatigue, Post traumatic stress disorder (PTSD), anxiety and depression.
3. One year after ICU discharge - the same as 3 months.

Survey instruments:

Pain - Brief Pain Inventory, Neuropathic Pain Syndrome Inventory, Pain diary QoL - SF 12, Sleep - General Sleep Disorder Scale Fatigue - Lee Fatigue Scale Anxiety and depression - Hospital Anxiety and Depression Scale PTSD - PTSS 10 Social Provision - Revised Social Provision Scale

ELIGIBILITY:
Inclusion Criteria:

* ICU stay longer than 48 h
* 18 years old or older
* Patients must write and understand Norwegian well.

Exclusion Criteria:

* Dying patients
* No acceptance form next of kind
* No concent from the patients
* Other that the researcher thinks should be excluded f. ex Patients with very bad prognosis
* Patients with low probability for self report after ICU stay

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in a Norwegian ICU. Medical and surgical patients, no thorasic surgery or trauma.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2010-05; Primary Completion 2018-04-30 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Do pain change over time in ICU survivors meassured with BPI and NPSI? | 1year after ICU discharge
  We will compare the results from 3 months with 1 year and look for differences.

SECONDARY OUTCOMES:
What is the relationship between patients self reported experience of pain and neurophysiological findings? | 3 months after ICU discharge
What is the relationship between patients self reported experience of pain and neurophysiological findings? | 1 year after ICU discharge
How are ICU survivors health related quality of life meassured with SF12? | 3 months after ICU discharge
How are ICU survivors health related quality of life meassured with SF 12? | 1 year after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Audun Stubhaug, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Langerud AK, Rustoen T, Smastuen MC, Kongsgaard U, Stubhaug A. Intensive care survivor-reported symptoms: a longitudinal study of survivors' symptoms. Nurs Crit Care. 2018 Jan;23(1):48-54. doi: 10.1111/nicc.12330. Epub 2017 Dec 15. PMID 29243344